CLINICAL TRIAL: NCT04742933
Title: A Head-to-Head Prospective Comparison of Diagnostic Accuracy of CCTA and Dynamic CT Perfusion in Patients With Prior PCI for the Diagnosis of Myocardial Ischemia as Defined by Invasive Flow and Pressure Indices - PACIFIC-III
Brief Title: CCTA and Dynamic CT Perfusion for the Diagnosis of Myocardial Ischemia in Patients With Coronary Stents
Acronym: PACIFIC-III
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Ibrahim Danad, MD, Principal Investigator, Amsterdam UMC, location VUmc
Other Study IDs: VUmc_2020-4973
Record Dates: First submitted 2021-02-02; First posted 2021-02-08 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Coronary Artery Disease
Keywords: Computed tomography angiography; Computed tomography Perfusion; FFR; Prior revascularization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 blood samples (21.5 Ml) for the PACIFIC 3 Biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: There is no intervention in this observational trial — There is no intervention in this observational trial

SUMMARY:
A single centre prospective trial in which patients with a prior PCI for stable CAD who are referred for invasive angiography will undergo state-of-the art CCTA and dynamic CT perfusion. Subsequently invasive FFR and iFR measurements will be routinely performed in each coronary vessel.

DETAILED DESCRIPTION:
Rationale: Recent development in computed tomography (CT) hardware have fulfilled the prerequisites for clinical CT myocardial perfusion imaging (CTP). Cardiac CT, has by means of coronary computed tomography angiography (CCTA) and novel techniques such as CTP the unique ability to provide information on both the anatomical and functional severity of coronary artery disease (CAD). However, diagnostic performance of these novel techniques when referenced by the clinical diagnostic standard, invasive fractional flow reserve (FFR) measurements, has scarcely been investigated in patients with a prior PCI.

Objective: To determine the diagnostic performance of CCTA and dynamic CTP for the diagnosis of myocardial ischemia using invasive coronary indices as the reference standard.

Study design: The study is a single-center prospective comparative trial in which all patients will undergo CCTA and dynamic CTP before invasive coronary angiography (ICA) in conjunction with invasive flow/pressure measurements.

Study population: Patients referred for a diagnostic ICA with a prior of PCI for stable CAD will be evaluated for inclusion in the study.

Main study parameters/endpoints: Hemodynamic significant CAD as defined by an FFR ≤0.80 / iFR < 0.90. Sensitivity, specificity, negative predictive value, positive predictive value and accuracy will be assessed for CCTA and dynamic CTP. In addition, this study will assess the prognostic value of CCTA and dynamic CTP in patients with a prior cardiac revascularization.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: A two day protocol will be completed after referral ensuring the diagnostic work-up of patients is not delayed. On day 1 patients will undergo CCTA and CTP. Then, on day 2, irrespective of CT results, patients will undergo ICA with invasive pressure measurements. The risks of CT are considered to be low. Patients are referred for a clinically indicated ICA and as such risks of the ICA are not deemed study-related. Future patients might benefit from the present study as combined anatomical information (CCTA) and functional information (dynamic CTP) might lead to a more judicious referral for ICA which leads to a reduction of exposure to invasive procedures such as ICA in combination with invasive pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* History of PCI for stable CAD
* Referred for a diagnostic ICA.
* Age above 30 years.

Exclusion Criteria:

* History of severe COPD or chronic asthma
* Pregnancy
* Renal failure (eGFR <30 mL/min)
* Use of sildenafil (Viagra) or dipyramidol (Persantin) that cannot be terminated
* Contra-indications for β-blockers
* Allergic reaction to iodized contrast
* Concurrent or prior (within last 30 days) participation in other research studies using investigational drugs
* Claustrophobia
* Significant co-morbidities
* Atrial fibrillation, second or third degree atrioventricular block
* Tachycardia
* Acute myocardial infarction
* History of CABG
* Heart failure
* Cardiomyopathies
* Previous radiation exposure in the diagnostic work-up
* Unable to give informed consent
* Indispensable follow-up with (serial) CT scans for non-cardiac related condition

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for a diagnostic ICA with a prior of PCI for stable CAD will be evaluated for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-25 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Dynamic CT-perfusion and CCTA for CAD | 3 years
  FFR will be used as a reference standard, the primary endpoint is an abnormal FFR =< 0.80. Diagnostic study using FFR as endpoun

SECONDARY OUTCOMES:
Major adverse cardiac events, cardiac death or repeat revascularization | 3 years
  The secondary endpoint is to assess the prognostic value of CT in patients with a prior history of PCI

CONTACTS AND LOCATIONS:
Overall Officials: Paul Knaapen, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc; Ibrahim Danad, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- Amsterdam UMC, location VUMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No